CLINICAL TRIAL: NCT04556851
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Trial of the Efficacy and Safety of HSK7653 as Monotherapy in Chinese Patients With Type 2 Diabetes
Brief Title: HSK7653 Treatment in Patients With Type 2 Diabetes Who Are Not Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK7653-301; CTR20201759 (Other: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK7653 10 mg (Experimental)
  Interventions: Drug: HSK7653 10 mg Q2W
- HSK7653 25 mg (Experimental)
  Interventions: Drug: HSK7653 25 mg Q2W
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK7653 10 mg Q2W — HSK7653 5 mg (2 tablets) and placebo 25 mg (1 tablet), Q2W, oral, week 1 to week 24; HSK7653 25 mg (1 tablet), Q2W, oral, week 25 to week 52.
  Arms: HSK7653 10 mg
Drug: HSK7653 25 mg Q2W — HSK7653 25 mg (1 tablet) and placebo 5 mg (2 tablets), Q2W, oral, week 1 to week 24; HSK7653 25 mg (1 tablet), Q2W, oral, week 25 to week 52.
  Arms: HSK7653 25 mg
Drug: Placebo — Placebo 25 mg (1 tablet) and placebo 5 mg (2 tablets), Q2W, oral, week 1 to week 24; HSK7653 25 mg (1 tablet), Q2W, oral, week 25 to week 52.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of HSK7653 (as monotherapy) compared with placebo after 24 weeks, and the safety (up to 52 weeks) of HSK7653 in Chinese patients with Type 2 diabetes who are insufficient glycaemic control with diet and exercise.

DETAILED DESCRIPTION:
The treatment period is composed of a 24-week double-blind period (week 1-24) and a 28-week open-label period (week 25-52). During the double-blind period, participants will receive 10 mg or 25 mg dose of HSK7653 and matching placebo, or placebo only. During the open-label period, all participants will receive 25 mg dose of HSK7653.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years, Male and female patients;
* Type 2 diabetes mellitus;
* Control the blood glucose level only with diet and exercise in last 8 weeks;
* Did not receive regular long-term medication of oral hypoglycemic drugs or insulin within 1 year prior to informed consent;
* HbA1c in the range of ≥7.5 to ≤11.0% at screening;
* FPG < 15 mmol/L at screening;
* BMI (Body Mass Index) in the range of ≥ 18.0 kg/m² to ≤ 35.0 kg/m² at screening.

Exclusion Criteria:

* Diabetic ketoacidosis, hyperglycemia hypertonic state, serious complications of diabetes, myocardial infarction, stroke within 6 months prior to informed consent;
* History of severe endocrine disease, uncured cancer, acute pancreatitis prior to informed consent;
* Current hemoglobinopathy, uncontrolled hypertension, serious nephropathy or hepatopathy prior to informed consent;
* Serious gastrointestinal disease within 2 weeks prior to informed consent;
* Serious infection, trauma and surgery within 3 months prior to informed consent;
* History of treatment with Dipeptidyl-Peptidase 4 (DPP-4) inhibitor, Glucose-dependent insulinotropic polypeptide (GIP) or Glucagon-like peptide-1 (GLP-1) receptor agonist;
* Treatment with drugs that affect glucose metabolism within 8 weeks prior to informed consent;
* Hemoglobin (HGB) < 10.0 g/dL(100 g/L);
* Alcohol abuse within 6 months or drug abuse history within 5 years prior to informed consent;
* Active infectious diseases;
* Participation in another trial with an investigational drug or instrument within 3 months prior to informed consent;
* Women who are nursing or pregnant, or subjects with birth plans;
* Contraindication for metformin;
* Other protocol-defined inclusion/exclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline at week 24 | Baseline and week 24
  Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24

SECONDARY OUTCOMES:
The Safety of HSK7653 at Week 24 and Week 52 | Baseline, week 24 and week 52
  Incidence of Treatment-Emergent Adverse Events over time (at week 24 and week 52)
Percentage of Patients With HbA1c <7.0% | Baseline, week 24 and week 52
Percentage of Patients With HbA1c <6.5% | Baseline, week 24 and week 52
FPG Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
2h-PPG Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Weight Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Fasting C-peptide Change From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Insulin Sensitivity Change (Calculated by HOMA-IS) From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Pancreatic β-cell function Change (Calculated by HOMA-β ) From Baseline at Week 24 and Week 52 | Baseline, week 24 and week 52
Percentage of Patients Required Use of Rescue Therapy or Dropout due to Hyperglycemia | Baseline, week 24 and week 52

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Zhujiang, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao L, Bian F, Pan T, Jiang H, Feng B, Jiang C, Sun J, Xiao J, Yan P, Ji L. Efficacy and safety of cofrogliptin once every 2 weeks in Chinese patients with type 2 diabetes: A randomized, double-blind, placebo-controlled, phase 3 trial. Diabetes Obes Metab. 2025 Jan;27(1):280-290. doi: 10.1111/dom.16014. Epub 2024 Oct 21. PMID 39434431